CLINICAL TRIAL: NCT06439602
Title: A Phase 3 Randomized, Double-blind, Multi-center, Placebo-controlled Study to Evaluate the Efficacy and Safety of AR882 in Participants With Gout
Brief Title: Phase 3 Evaluation of Efficacy and Safety of AR882 in Gout Patients (AR882-302)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR882-302
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Gout; Arthritis, Gouty; Hyperuricemia; Gout Chronic
MeSH Terms: conditions — Gout; Arthritis, Gouty; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AR882 50 mg (Experimental): AR882 50 mg taken once daily for 12 months
  Interventions: Drug: AR882 50 mg
- AR882 75 mg (Experimental): AR882 75 mg taken once daily for 12 months
  Interventions: Drug: AR882 75 mg
- Placebo (Placebo Comparator): AR882 matching placebo taken once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR882 50 mg — Solid Oral Capsule
  Arms: AR882 50 mg
Drug: AR882 75 mg — Solid Oral Capsule
  Arms: AR882 75 mg
Drug: Placebo — Matching Solid Oral Capsule Placebo
  Arms: Placebo

SUMMARY:
This study will assess the serum uric acid lowering effect and safety of AR882 in gout patients at two doses compared to placebo over 12 months

ELIGIBILITY:
Inclusion Criteria:

* History of gout
* Occurrence of ≥ 2 self-reported gout flares in the last 12 months
* Body weight no less than 50 kg
* Patients who are NOT on approved urate-lowering therapy (ULT) must have sUA ≥ 7 mg/dL
* Patients who are on medically appropriate ULT must have sUA > 6 mg/dL
* Serum creatinine must be < 3.0 mg/dL and estimated CLcr ≥ 30 mL/min

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* Pregnant or breastfeeding
* History of symptomatic kidney stones within the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 6 mg/dL at month 6 | 24 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL at month 6

SECONDARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 6 mg/dL from the end of month 9 to the end of month 12 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL for the 3-month period from the end of month 9 to the end of month 12
No gout flares from the end of month 9 to the end of month 12 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with no gout flares for the 3-month period from the end of month 9 to the end of month 12
Change in tophus burden by month 12 | 48 weeks
  Comparison of the treatment groups for the proportion of patients who experience a complete response, marked or partial response, of at least 1 target tophus at Month 12, with no evidence of disease progression (no new tophus or single tophus showing progression) and patients with no new tophi formation at month 12 as determined using the computer-assisted photographic evaluation in rheumatology (CAPER) method
Incidence of Adverse Events | 56 weeks
  Treatment Emergent Adverse Events and Serious Adverse Event incidence

CONTACTS AND LOCATIONS:
Overall Officials: Robert Keenan, MD, Study Director — Arthrosi Therapeutics, Inc.
Locations (68):
- United States (52):
  - Arthrosi Investigative Site (106), Foley, Alabama
  - Arthrosi Investigative Site (139), Anchorage, Alaska
  - Arthrosi Investigative Site (160), Peoria, Arizona
  - Arthrosi Investigative Site (112), Phoenix, Arizona
  - Arthrosi Investigative Site (114), Tempe, Arizona
  - Arthrosi Investigative Site (131), El Cajon, California
  - Arthrosi Investigative Site (117), Encinitas, California
  - Arthrosi Investigative Site (138), Rancho Cucamonga, California
  - Arthrosi Investigative Site (161), Valencia, California
  - Arthrosi Investigative Site (101), Aurora, Colorado
  - Arthrosi Investigative Site (149), Clearwater, Florida
  - Arthrosi Investigative Site (115), Coral Gables, Florida
  - Arthrosi Investigative Site (128), DeLand, Florida
  - Arthrosi Investigative Site (102), Hollywood, Florida
  - Arthrosi Investigative Site (156), Maitland, Florida
  - Arthrosi Investigative Site (103), Miami, Florida
  - Arthrosi Investigative Site (157), Palmetto Bay, Florida
  - Arthrosi Investigative Site (151), Winter Haven, Florida
  - Arthrosi Investigative Site (164), Atlanta, Georgia
  - Arthrosi Investigative Site (162), Lilburn, Georgia
  - Arthrosi Investigative Site (133), Boise, Idaho
  - Arthrosi Investigative Site (122), River Forest, Illinois
  - Arthrosi Investigative Site (154), Wichita, Kansas
  - Arthrosi Investigative Site (144), New Orleans, Louisiana
  - Arthrosi Investigative Site (150), Hagerstown, Maryland
  - Arthrosi Investigative Site (121), Ann Arbor, Michigan
  - Arthrosi Investigative Site (105), Detroit, Michigan
  - Arthrosi Investigative Site (153), Olive Branch, Mississippi
  - Arthrosi Investigative Site (119), Kansas City, Missouri
  - Arthrosi Investigative Site (158), Brooklyn, New York
  - Arthrosi Investigative Site (137), Greensboro, North Carolina
  - Arthrosi Investigative Site (140), Shelby, North Carolina
  - Arthrosi Investigative Site (130), Wilmington, North Carolina
  - Arthrosi Investigative Site (148), Cleveland, Ohio
  - Arthrosi Investigative Site (146), Dayton, Ohio
  - Arthrosi Investigative Site (120), Hatboro, Pennsylvania
  - Arthrosi Investigative Site (147), Myrtle Beach, South Carolina
  - Arthrosi Investigative Site (132), Rapid City, South Dakota
  - Arthrosi Investigative Site (110), Amarillo, Texas
  - Arthrosi Investigative Site (104), Dallas, Texas
  - Arthrosi Investigative Site (116), Graham, Texas
  - Arthrosi Investigative Site (126), Lake Jackson, Texas
  - Arthrosi Investigative Site (136), Missouri City, Texas
  - Arthrosi Investigative Site (129), Plano, Texas
  - Arthrosi Investigative Site (127), Round Rock, Texas
  - Arthrosi Investigative Site (107), Tomball, Texas
  - Arthrosi Investigative Site (124), Tomball, Texas
  - Arthrosi Investigative Site (142), Bountiful, Utah
  - Arthrosi Investigative Site (145), Ogden, Utah
  - Arthrosi Investigative Site (111), Hampton, Virginia
  - Arthrosi Investigative Site (118), Hampton, Virginia
  - Arthrosi Investigative Site (134), Winchester, Virginia
- Australia (2):
  - Arthrosi Investigative Site (202), Botany, New South Wales
  - Arthrosi Investigative Site (200), Camberwell, Victoria
- Hong Kong (2):
  - Arthrosi Investigative Site (500), Hong Kong, Central
  - Arthrosi Investigative Site (501), Hong Kong, Hong Kong Island
- New Zealand (5):
  - Arthrosi Investigative Site (300), Auckland, Auckland
  - Arthrosi Investigative Site (304), Hamilton, Hamilton
  - Arthrosi Investigative Site (302), Auckland, New Zealand
  - Arthrosi Investigative Site (303), Nelson, New Zealand
  - Arthrosi Investigative Site (301), Rotorua, New Zealand
- Taiwan (7):
  - Arthrosi Investigative Site (405), Hualien City, Taiwan
  - Arthrosi Investigative Site (404), Kaohsiung City, Taiwan
  - Arthrosi Investigative Site (400), Taipei, Taiwan
  - Arthrosi Investigative Site (403), Taipei, Taiwan
  - Arthrosi Investigative Site (401), Taoyuan, Taiwan
  - Arthrosi Investigative Site (406), Kaohsiung City
  - Arthrosi Investigative Site (402), Taichung

IPD SHARING:
Plan to Share IPD: No